CLINICAL TRIAL: NCT07407049
Title: Comparison of Early Postoperative Visual Acuity Between Intracapsular and Supracapsular Phacoemulsification: A Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025KYPJ174
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supracapsular Phacoemulsification (Active Comparator)
  Interventions: Procedure: Supracapsular Phacoemulsification
- Intracapsular Phacoemulsification (Experimental)
  Interventions: Procedure: Intracapsular Phacoemulsification

INTERVENTIONS:
Procedure: Supracapsular Phacoemulsification — During phacoemulsification, real-time imaging of the anterior segment was performed using SS-iOCT (Tupai, China), but the surgeon was not able to view the images. The surgeon was instructed to proceed with phacoemulsification as per routine, using phaco energy (i.e., level 3). All other surgical steps were identical to conventional surgery.
  Arms: Supracapsular Phacoemulsification
Procedure: Intracapsular Phacoemulsification — During phacoemulsification, real-time imaging of the anterior segment was performed using SS-iOCT (Tupai, China). The surgeon was required to confirm under SS-iOCT guidance that the phaco tip was located within the capsular bag (as judged by two observers not involved in the surgery) before applying phaco energy (i.e., level 3). All other surgical steps were identical to conventional surgery.
  Arms: Intracapsular Phacoemulsification

SUMMARY:
Cataracts are the leading cause of blindness worldwide, and phacoemulsification combined with intraocular lens implantation has become the most mainstream surgical approach. With advancements in surgical techniques and equipment, this procedure has evolved from a simple vision-restoring surgery into the era of refractive surgery. Patients now have higher expectations for postoperative visual quality, particularly the recovery of early vision, which directly impacts their satisfaction. Intraoperative surgical details have a direct influence on postoperative visual acuity.

Thanks to intraoperative optical coherence tomography (iOCT) technology, surgeons have gradually recognized that factors such as surgical incisions and intraoperative anterior chamber collapse can affect the survival of corneal endothelial cells after surgery, which is directly related to early postoperative vision and patient satisfaction. Swept-source intraoperative OCT (SS-iOCT) has further improved imaging range and clarity, helping us discover that the depth of intraoperative ultrasound energy use (such as cumulative dissipated energy) correlates with postoperative corneal endothelial cell loss. This suggests that compared to performing phacoemulsification at the capsular opening plane or in the anterior chamber, intracapsular phacoemulsification may reduce postoperative corneal endothelial cell loss, potentially leading to better early postoperative vision, which is crucial for patient satisfaction. However, evidence is still lacking.

Therefore, this study aims to compare the effects of intracapsular versus extracapsular phacoemulsification on early postoperative vision, as well as long-term visual acuity, corneal endothelial cells, corneal changes, and the incidence of intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years and ≤ 90 years
* Able to cooperate with preoperative examinations
* At least one eye meets the study eye criteria
* Has the capacity and willingness to provide informed consent
* Age-related cataract
* Nuclear opacity (N) graded ≥4 according to the Lens Opacities Classification System III (LOCS III)
* Scheduled for phacoemulsification with intraocular lens implantation
* Pupil size ≥6 mm after dilation
* Corneal endothelial cell density ≥1500 cells/mm²

Exclusion Criteria:

* Considered unsuitable by the investigator for participation in this clinical trial for other reasons (e.g., unstable systemic condition, uncontrolled blood pressure/blood glucose, severe cardiovascular disease, renal disease, etc.)
* Blood pressure > 180/110 mmHg (systolic >180 mmHg or diastolic >110 mmHg). Patients may be considered for inclusion if blood pressure can be controlled below these thresholds with medication.
* History of myocardial infarction or other cardiac disease requiring hospitalization, cerebral infarction, transient ischemic attack, or acute heart failure within 4 months prior to enrollment.
* Women with childbearing potential (i.e., currently pregnant, breastfeeding, or planning to become pregnant within the next 2 years). Women of childbearing potential should be asked about the possibility of pregnancy, and the investigator will determine when a pregnancy test is necessary.
* Currently participating in another clinical trial
* History of ocular trauma or surgery
* Presence of other ocular diseases (e.g., glaucoma, diabetic retinopathy)
* Other ocular factors that may complicate surgery (e.g., small pupil, shallow anterior chamber)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The best-corrected distance visual acuity at 1 day postoperatively. | 1 day postoperatively
  It was evaluated using the ETDRS visual acuity chart by a masked optometrist, with the examination procedure following the standard ETDRS visual acuity testing protocol, and the unit of measurement was logMAR.

SECONDARY OUTCOMES:
Coefficient of variation of corneal endothelial cell size | Post-operative day 1, week 1, month 1, month 3, month 6
The percentage loss of central corneal endothelial cell density compared to the preoperative baseline at post-operative day 1 and post-operative | 1 day and 1 month postoperatively
Percentage of hexagonal cells | Post-operative day 1, week 1, month 1, month 3, month 6
Central corneal thickness | Post-operative day 1, week 1, month 1, month 3, month 6
Corneal endothelial cell density | Post-operative day 1, week 1, month 1, month 3, month 6
The best-corrected distance visual acuity at other time frame | Post-operative week 1, month 1, month 3, month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China